CLINICAL TRIAL: NCT02465632
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Glenmark Generics, Ltd) to the Marketed Product BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5% (Valeant Pharmaceuticals, US) in the Treatment of Acne Vulgaris.
Brief Title: To Study Generic Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Glenmark Generics, Ltd) in the Treatment of Acne Vulgaris.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLK-1403
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2015-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel (Experimental): apply a thin layer of gel to the face
  Interventions: Drug: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
- BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5% (Active Comparator): apply a thin layer of the gel to the face
  Interventions: Drug: BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%
- Placebo topical gel (Placebo Comparator): apply a thin layer of the gel to the face
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
  Arms: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
Drug: BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%
  Arms: BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%
Drug: Placebo
  Arms: Placebo topical gel

SUMMARY:
This is a randomized, double-blind, multiple-site, placebo-controlled, parallel-group study, designed to compare the efficacy and safety of generic Clindamycin 1%/ Benzoyl peroxide 5% topical gel (Glenmark Generics, Ltd), and the marketed product BenzaClin® Topical Gel, Clindamycin 1%/ Benzoyl peroxide 5% (Valeant Pharmaceuticals, US) in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, ≥12 and ≤40 years of age with a clinical diagnosis of acne vulgaris.
2. Have facial acne with: ≥20 facial inflammatory lesions (papules and pustules) and ≥25 non-inflammatory lesions (open and closed comedones), and ≤2 nodulocystic lesions (nodules and cysts) and have an IGA score of 2, 3 or 4.

Exclusion Criteria:

1. Subject has more than 2 facial nodular lesions; any nodules present will be documented but not included in the inflammatory lesion count for analysis.
2. Subject has active cystic acne.
3. Subject has acne conglobata.
4. Subjects with excessive facial hair such as beards, sideburns, moustaches, etc. that would interfere with the diagnosis or assessment of acne.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1100 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh V Deshpande, Study Director — Glenmark Pharmaceuticals Ltd
Locations (15):
- United States (13):
  - Glenmark Investigational Site 13, Anaheim, California
  - Glenmark Investigational Site 6, Long Beach, California
  - Glenmark Investigational Site 15, Los Angeles, California
  - Glenmark Investigational Site12, West Covina, California
  - Glenmark Investigational Site 4, Brandon, Florida
  - Glenmark Investigational Site 1, Miami, Florida
  - Glenmark Investigational Site 8, Miami, Florida
  - Glenmark Investigational Site 9, Miramar, Florida
  - Glenmark Investigational Site 2, St. Petersburg, Florida
  - Glenmark Investigational Site 5, Louisville, Kentucky
  - Glenmark Investigational Site7, Upper Saint Clair, Pennsylvania
  - Glenmark Investigational Site 14, Greenville, South Carolina
  - Glenmark Investigational Site 3, Nashville, Tennessee
- Belize (2):
  - Glenmark Investigational Site 10, Belize City
  - Glenmark Investigational Site 11, Belize City

RESULTS

PARTICIPANT FLOW:
Groups:
- Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel: Test: A thin layer of gel was applied to the entire affected areas on the face twice a day.
- BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%: Reference: A thin layer of gel was applied to the entire affected areas on the face twice a day.
- Placebo Topical Gel: Placebo: A thin layer of gel was applied to the entire affected areas on the face twice a day.
Period: Overall Study
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel | BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5% | Placebo Topical Gel
Started | 440 | 440 | 220
Completed | 409 | 417 | 203
Not Completed | 31 | 23 | 17

BASELINE CHARACTERISTICS:
Population: A total of 1100 subjects were randomized in the study; of these 27 subjects did not received the dose (Test=8, Reference=10, Placebo=9) and were excluded from the safety population randomized. Therefore the overall number of subjects in the Baseline Participants module is not consistent with any of the rows of the Participant Flow module.
Groups:
- Test: Test: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
- Reference: Reference: BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%
- Placebo: Placebo: Placebo topical gel
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 432 | 430 | 211 | 1073
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (7.7) | 22.3 (7.6) | 22.6 (7.5) | 22.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 259 | 127 | 660
  Male | 158 | 171 | 84 | 413

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in the Number of Inflamed Lesions (Papules/Pustules)
Description: The number of inflammatory lesions (papules and pustules) count between the treatment groups were estimated.
Time Frame: Baseline and 10 Weeks
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Test: Clindamycin and Benzoyl Peroxide Gel, 1%/5%
- Reference: BenzaClin® Topical Gel: Clindamycin and Benzoyl Peroxide Gel, 1%/5%
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 362 | 368 | 176
percentage change from baseline | 72.3 (25.2) | 71.1 (26.7) | 39.1 (31.4)

2. Primary Outcome: Mean Percent Change in the Number of Non-inflamed Lesions (Open and Closed Comedones)
Description: The number of non-inflamed lesions (open and closed comedones) count between treatment groups were estimated.
Time Frame: Baseline and 10 Weeks
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 362 | 368 | 176
Percentage change from baseline | 64.5 (24.7) | 63.3 (26.2) | 30.9 (28.5)

ADVERSE EVENTS:
Description: A total of 1100 subjects were randomized in the study; of these 27 subjects did not received the dose (Test=8, Reference=10, Placebo=9) and were excluded from the safety population randomized. Therefore the total number of Participants at risk is not consistent with any of the rows of the Participant Flow module.
Groups:
- Test: Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel
- Reference: BenzaClin® Topical Gel, Clindamycin 1%/Benzoyl Peroxide 5%
- Placebo: Placebo topical gel
Arm/Group | Test | Reference | Placebo
Serious Adverse Events (participants affected / at risk) | 0/432 | 0/430 | 0/211
Other Adverse Events (participants affected / at risk) | 0/432 | 0/430 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the agreement, Sponsor reserves the right for publishing trial results and the Investigator cannot publish without written consent from the Sponsor.